CLINICAL TRIAL: NCT02651090
Title: Evaluation of Suspected Liver Pathology in Patients With Contraindications for Contrast Enhanced Computed Tomography and/or Magnetic Resonance Imaging Using Sonazoid
Brief Title: Evaluation of Suspected Liver Pathology in Patients With Contraindications for Contrast Enhanced CT and/or MRI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated study before enrollment Sponsor terminated study before enrollment
Sponsor: Northeastern Ohio Radiology Research and Education Fund (Other)
Responsible Party: Principal Investigator, Richard G. Barr MD, PhD, Medical Director, Northeastern Ohio Radiology Research and Education Fund
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SONA1
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Liver Metastasis; Liver Mass
Keywords: contraindication for CECT; contraindication for CEMRI; liver pathology; renal failure; contrast enhanced ultrasound; sonazoid
MeSH Terms: conditions — Renal Insufficiency | interventions — Sonazoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sonazoid (Experimental): treatment arm with sonazoid
  Interventions: Drug: Sonazoid

INTERVENTIONS:
Drug: Sonazoid — Comparison of Sonazoid enhanced ultrasound to non enhanced CT
  Other Names: NC100100

SUMMARY:
Patients with renal failure or other reason for contraindication for contrast enhanced computed tomography (CECT) or contrast enhanced magnetic resonance imaging (CEMRI) with suspected liver pathology will be evaluated with Sonazoid enhanced Ultrasound

DETAILED DESCRIPTION:
Patients with a diagnosis of cancer or high probability of cancer (any primary) who have contraindications for a contrast enhanced Computed Tomography or Magnetic Resonance Image will be asked to participate in this study. Patients will be both male and female and be >18 years old. Contraindications for computer tomography (CT) or magnetic resonance imaging (MRI) would include, but not limited to:

1. Creatinine clearance of <60 mg/dl
2. Allergy to iodinated contrast or gadolinium based contrast agents
3. History of adverse event with CT or MRI contrast

Up to 100 patients will be enrolled over a two year period.

Statistical justification for sample size Assuming that a non-enhanced CT will detect and characterize metastatic disease correctly 60% of the time (2) and that Contrast enhanced ultrasound (CEUS) will detect and characterize metastatic disease correctly 90% of the time (3,4), there will be a 100% chance of a significant difference at a one-sided 0.05 significance level using the Fisher Exact Test.

CT and MRI Patient will receive the non-contrast CT or MRI that would be ordered as routine stating or follow-up of the patient. At a minimum 5mm contiguous axial slices will be obtained with CT and T1-weighted, T2-weighted, in-phase and out of phase imaging will be performed on MRI with a minimum slice thickness of 5mm. Each lesion noted within the liver will be measured in two dimensions and recorded. The lesion will be classified on a scale of 1 - 5 regarding the probability of benignity or malignancy of the lesion. If a diagnosis can be made the diagnosis will be documented The location of the lesion will be documented on a Couinaud diagram.

CEUS-Contrast specific software optimized for Sonazoid will be used or both vascular and Kupffer phase imaging. The focus will be set below the lesion of interest for vascular phase imaging and at 4-8 cm for the left lobe and 8-10 cm for the right lobe for Kupffer phase imaging. The lesion of interest was imaged from 15 seconds before injection to 1 minute after injection (vascular phase imaging). No further scanning will be performed until the Kupffer phase imaging, which will begun 10 minutes after the injection.

The patient will receive the following ultrasound imaging:

1. Standard B-mode and color-Doppler imaging. Elastography may be added at PI's discretion.
2. A 20g IV will be placed in an antecubital vein
3. Low MI scan will be used in the vascular phase.
4. An intermediate MI scan will be used after at least a 10 minute delay to perform the Kupffer scan
5. If a lesion is identified on the Kupffer scan which is not characterized by the without exam the patient will have a complete evaluation of the vascular phase a second injection may be used.

Each lesion noted within the liver will be measured in two dimensions and recorded. The lesion will be classified on a scale of 1 - 5 regarding the probability of benignity or malignancy of the lesion. If a diagnosis can be made the diagnosis will be documented. The location of the lesion will be documented on a Couinaud Diagram.

The gold standard will be either

1. characteristic enhancement pattern (hemangioma, benign)
2. lesion biopsy
3. growth of the lesion over a 6 month period of time (malignant)

Data Analysis

For assessment of characterization efficacy the McNemar test will be used to compare the rates of correct diagnosis for lesions on unenhanced ultrasound, CEUS and unenhanced CT or MRI. For assessment of detection efficacy, Wilcoxon's signed rank test will be used to compare the lesion detection rates obtained with unenhanced ultrasound, CEUS, and unenhanced CT or MRI. For all tests, p<0.05 will be considered a statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of cancer or a high probability of having cancer but not yet diagnosed who have a contraindication to a contrast CT or MRI
2. Age >18 years
3. No know allergies to Sonozoid
4. Ability to give informed consent

Exclusion Criteria:

1. No IV access
2. Inability to give informed consent
3. Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The detection rate of Sonozoid enhanced US for focal liver lesions in patients unable to have a contrast enhanced CT or MRI compared to unenhanced CT or MRI | 2 years
  Determination of the liver lesion detection rate of Sonozoid
Focal liver characterization as benign, Indeterminate, or malignant by Sonozoid enhanced ultrasound in compared to unenhanced CT or MRI. | 2 years
  Determine the accuracy of liver lesion characterization by Sonozoid

SECONDARY OUTCOMES:
Title: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0 | 2 years
  Evaluate the Adverse event rate using Sonozoid